CLINICAL TRIAL: NCT03292913
Title: Positive Health Check Evaluation Trial
Acronym: (PHC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1U18PS004967-01 (NIH)
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Results first posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Human Immunodeficiency Virus (HIV) Positive
Keywords: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — HIV Seropositivity; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receives the Positive Health Check intervention plus standard of care
  Interventions: Behavioral: Positive Health Check
- Control Group (Other): Receives standard of care
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Positive Health Check — Positive Health Check (PHC) is an online intervention that delivers tailored evidence-based prevention messages to human immunodeficiency virus (HIV) positive patients through a series of brief interactive videos designed to simulate a conversation with an human immunodeficiency virus (HIV) primary care provider.
  Arms: Intervention Group
Behavioral: Standard of Care — Standard of care for patients with human immunodeficiency virus (HIV) (this includes standard of care practices around antiretroviral therapy (ART) initiation, adherence and retention)
  Arms: Control Group

SUMMARY:
The purpose of the study is to evaluate the effect of Positive Health Check (PHC), an online intervention that delivers tailored, evidence-based prevention messages to HIV positive patients, on improving clinical outcomes and retention in care of people who are HIV positive and have unsuppressed viral loads. The costs and processes of implementation will also be assessed to inform future dissemination.

DETAILED DESCRIPTION:
The Positive Health Check (PHC) Evaluation Trial uses a randomized trial to test if a brief web-based counseling intervention can improve clinical outcomes among people living with human immunodeficiency virus (HIV). The study will also assess implementation processes, collect data to determine cost effectiveness, and document the standard of care in each clinic. The study will take place in four locations including Atlanta Veterans Affairs (VA) Medical Center (Atlanta, GA), Hillsborough County Health Department (Tampa, FL), Rutgers Infectious Disease Practice (Newark, NJ) and Crescent Care (New Orleans, LA). The objectives of the PHC Evaluation Trial are four-fold: Objective 1) Implement a randomized trial to test if the PHC intervention improves clinical health outcomes, specifically viral load suppression and retention in care. While Positive Health Check (PHC) is designed to improve antiretroviral therapy (ART) initiation, ART adherence and retention in care as well as reduce unprotected sex and promote safe injection practices, the primary outcome on which the trial is powered is viral suppression; Objective 2) Conduct an implementation evaluation to determine effective implementation strategies and integration of Positive Health Check (PHC) into human immunodeficiency virus (HIV) primary care clinics; Objective 3) Collect and document data on the cost of the PHC intervention implementation; Objective 4) Document the standard of care at each participating site. Positive Health Check (PHC) is a web-based intervention that delivers tailored evidence-based prevention messages to human immunodeficiency virus (HIV) positive patients through a series of brief interactive videos designed to simulate a conversation with an human immunodeficiency virus (HIV) primary care provider. Web-based interventions have been shown to be effective in improving adherence and reducing sexual risk. Eligible patients, who use the intervention, are given a tablet with a privacy screen, a set of headphones, a unique login identification (ID) and will be prompted to create their own private password. Once logged in, the intervention guides a patient through tailored messaging from a video doctor on patient-selected topics including treatment initiation or adherence, retention in care, sexual risk reduction, pregnancy, and intravenous drug use. Throughout the intervention patients answer tailoring questions about themselves and based on their answers, are given tailored messages from their chosen video doctor. Positive Health Check (PHC) is designed to facilitate patient-provider communication on these topics. In the intervention, patients can select which questions they have for their doctor on the topics covered and which health promotion strategies they want to practice before their next visit. The questions and chosen health promotion strategies ("tips") automatically populate to a handout which is given to the patient after logging off. Patients also have access to another module that provides other information about human immunodeficiency virus (HIV) management, how to prevent transmission, and living a healthy lifestyle while being human immunodeficiency virus (HIV) positive. The intervention will be considered implemented with fidelity if a patient completes the intervention in the clinic before or after seeing their primary care provider, or before or after a blood draw or ancillary appointment in advance of their appointment with their clinical provider. A patient may also begin the intervention in the clinic and complete it after the appointment or at home within 21 days. Evaluation of the intervention will include comparisons of the intervention and control arms on the primary outcome using data abstracted via electronic medical records, with the 12- month viral load value considered the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Diagnosed with human immunodeficiency virus (HIV);
3. English-speaking;
4. Attending one of the four clinical sites;
5. Meet at least one of the following: a) Most recent viral load lab result of ≥ 200 copies/mL, b) Attended an initial human immunodeficiency virus human immunodeficiency virus (HIV) appointment with a provider at one of the four sites within the past 12 months; c) Out of care (last attended appointment at the clinic was more than 12 months ago);
6. Not involved in any other intervention that would bias outcome assessment,
7. Deemed mentally competent and able to engage with the intervention.

Exclusion Criteria:

1. Under 18 years of age;
2. Human immunodeficiency virus (HIV) negative;
3. Does not speak English;
4. Does not attend one of the four clinical sites for (HIV) primary care;
5. Meets all of the following: a) Most recent viral load lab result of < 200 copies/mL, b) Did not attend an initial human immunodeficiency virus (HIV) appointment with a provider at one of the four sites within the past 12 months, c) Last attended appointment at the clinic was less than 12 months ago)
6. Involved in an intervention that would bias outcome assessment;
7. Deemed mentally incompetent to engage with the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Lewis, PhD, Principal Investigator — RTI International
Locations (4):
- United States (4):
  - Hillsborough County Health Department, Tampa, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Crescent Care, New Orleans, Louisiana
  - Rutgers Infectious Disease Practice, Newark, New Jersey

REFERENCES:
- [Derived] Lewis MA, Harshbarger C, Bann C, Marconi VC, Somboonwit C, Piazza MD, Swaminathan S, Burrus O, Galindo C, Borkowf CB, Marks G, Karns S, Zulkiewicz B, Ortiz A, Abdallah I, Garner BR, Courtenay-Quirk C; Positive Health Check Study Team. Effectiveness of an Interactive, Highly Tailored "Video Doctor" Intervention to Suppress Viral Load and Retain Patients With HIV in Clinical Care: A Randomized Clinical Trial. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):58-67. doi: 10.1097/QAI.0000000000003045. Epub 2022 Jun 27. PMID 35972854

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Receives the Positive Health Check intervention plus standard of care
  Positive Health Check: PHC is an online intervention that delivers tailored evidence-based prevention messages to HIV positive patients through a series of brief interactive videos designed to simulate a conversation with an HIV primary care provider.
- Control Group: Receives standard of care
  Standard of Care: Standard of care for patients with HIV (this includes standard of care practices around ART initiation, adherence and retention)
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 397 | 402
Completed | 315 | 314
Not Completed | 82 | 88
Not completed — Death | 9 | 3
Not completed — Lost to Follow-up | 49 | 49
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Clinic closed due to COVID | 22 | 36

BASELINE CHARACTERISTICS:
Population: One of the 397 participants in the Positive Health Check and Standard of Care group and one of the 402 participants in the Standard of Care group were missing data for age because it was not included in their patient charts.
Groups:
- Intervention Group: Positive Health Check and Standard of Care
  Participants with HIV diagnosis received Positive Health Check intervention and standard of care
- Control Group: Standard of care
  Participants with HIV diagnosis received standard of care only
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 397 | 402 | 799
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 participants, 1 from each group did not declare their age.
  Participants
    Participants: number analyzed (Participants) | 396 | 401 | 797
    Participants: <=18 years | 0 | 0 | 0
    Participants: Between 18 and 65 years | 376 | 383 | 759
    Participants: >=65 years | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One of the 397 participants in the Positive Health Check and Standard of Care group and one of the 402 participants in the Standard of Care group were missing data for age because it was not included in their patient charts.
  years
    number analyzed (Participants) | 396 | 401 | 797
    (all) | 45.4 (13.0) | 44.5 (12.6) | 44.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant did not declare gender/sex
  Participants
    Participants: number analyzed (Participants) | 397 | 401 | 798
    Participants: Female | 303 | 306 | 609
    Participants: Male | 94 | 95 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 32 | 63
  Not Hispanic or Latino | 359 | 365 | 724
  Unknown or Not Reported | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 299 | 301 | 600
  White | 85 | 88 | 173
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants] — All participants data were included in the trial data that was analyzed regardless of the missing demographics data.
  participants
    United States | 397 | 402 | 799

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Load Suppression
Description: Viral load suppression was defined as having viral load < 200 copies/mL by the end of each participant's 12 months of follow-up assessment (with a window from start of 10 months through the end of 16 months post-randomization to accommodate timing of clinical visits).
Time Frame: Targeted time frame is 12 months post-randomization with a possible range of 10-16 months to account for variable timing of clinic visits.
Population: All participants with a viral load measurement at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Positive Health Check intervention plus standard of care
- Control Group: Standard of care only
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 368 | 372
Participants | 210 | 213
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Outcome measure for this analysis is viral load suppression. A priori threshold for statistical significance is p-value less than 0.05; Test type: Superiority; p = 0.220, Mixed Models Analysis; Risk ratio is adjusted for sex, age, race, site, viral load suppression at baseline, and new to care; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.96 to 1.21]

2. Secondary Outcome: Number of Participants Retained in Care at 12-month Follow up
Description: Retention in care is a patient defined as having at least one visit in each 6-month period within 12 months post-randomization separated by at least two months.
Time Frame: Up to 12 months post randomization
Population: All participants
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Participants with HIV diagnosis who received Positive Health Check intervention plus standard of care
- Control Group: Patients with HIV diagnosis who received standard of care only
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 397 | 402
Participants | 257 | 247
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Outcome measure for this analysis is retention in care. A priori threshold for statistical significance is p-value less than 0.05; Test type: Superiority; p = 0.481, Mixed Models Analysis; Risk ratio is adjusted for sex, age, race, site, and new to care; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.94 to 1.15]

3. Secondary Outcome: Retention in Care
Description: A 6-month visit gap was defined as having at least 189 days between two sequentially kept visits, post-randomization.
Time Frame: 12 months of randomization
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: Participants with human immunodeficiency virus (HIV) diagnosis who received Positive Health Check intervention plus standard of care
- Control Group: Patients with human immunodeficiency virus (HIV) diagnosis who received standard of care only
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 397 | 402
Participants | 113 | 164
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Outcome measure for this analysis is a 6-month visit gap defined ashaving at least 189 days between two sequentially kept visits, post-randomization. A priori threshold for statistical significance is p-value less than 0.05; Test type: Superiority; p = 0.093, Mixed Models Analysis; Risk ratio is adjusted for sex, age, race, site, and new to care; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.72 to 1.03]

ADVERSE EVENTS:
Time Frame: Baseline to 12 months post randomization
Description: Each death was reviewed by the respective site's study Institutional Review Board (IRB) and deemed not related with the trial.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 9/397 | 3/402
Serious Adverse Events (participants affected / at risk) | 0/397 | 0/402
Other Adverse Events (participants affected / at risk) | 0/397 | 0/402

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03292913/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03292913/SAP_001.pdf
  • Informed Consent Form (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03292913/ICF_002.pdf